CLINICAL TRIAL: NCT05607576
Title: Accuracy of Dexcom G6 After Radiation Exposure-A Cross Sectional and Longitudinal Analysis
Brief Title: Dexcom G6 for Total Pancreatectomy With Islet Autotransplantation (TPIAT) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Elder (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Deborah Elder, ASSOCIATE PROFESSOR, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0838
Record Dates: First submitted 2022-07-19; First posted 2022-11-07 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
Keywords: Dexcom G6
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: This study is not blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uncovered (Experimental): Dexcom G6 CGM will be uncovered during standard of care radiologic procedures.
  Interventions: Other: Uncovered CGM during radiologic procedures

INTERVENTIONS:
Other: Uncovered CGM during radiologic procedures — Dexcom G6 CGM will not be covered during radiologic procedures.

SUMMARY:
A single-center prospective trial on the effects of standard of care radiation exposure on the Dexcom G6 continuous glucose monitoring (CGM) device.

DETAILED DESCRIPTION:
To determine if standard of care radiation exposure longitudinally effects the accuracy and precision of the G6 transmitter in the post TPIAT in-patient population.

Reduce burden for patients to remove and waste a functional and expensive Dexcom G6 CGM for radiologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Planned TPIAT at CCHMC
* Staying in-patient at CCHMC post TPIAT
* Planned to receive a Dexcom G6 CGM

Exclusion Criteria:

• Hemo- or peritoneal dialysis

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deb Elder, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share any individual Participant data. We will be publishing aggregate data.

REFERENCES:
- [Result] Tellez S, Hornung L, Smith E, Trout A, Brady S, Lowe C, Courter J, Abu-El-Haija M, Elder D. Real-World Accuracy of a Continuous Glucose Monitoring System after Radiologic Exposure. Pediatr Diabetes. 2024 Aug 7;2024:2210509. doi: 10.1155/2024/2210509. eCollection 2024. PMID 40302953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uncovered
Started | 18
Completed | 14
Not Completed | 4
Not completed — immediate sensor error | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: 14 participants were enrolled and completed the study.
Arm/Group | Uncovered
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
BMI percentile [Mean (Inter-Quartile Range); unit: Percentile] | 79.4 [46.1 to 98.2]
Insurance [Count of Participants; unit: Participants]
  Private | 8
  Medicaid | 5
  Private and Medicaid | 1

OUTCOME MEASURES:

1. Primary Outcome: Dexcom G6 Accuracy Post Radiation Exposure by Clark Error Analysis (Zone A and B %)
Description: Blood Glucose levels (mg/dL) obtained by the Dexcom G6 sensor and transmitter compared to blood glucose levels (mg/dL) obtained by a handheld glucometer until the transmitter is changed. The Clarke Error Grid Analysis method was used to compare absolute values. Accuracy reported as percentage of comparators in Zone A and B.
Time Frame: 3 months
Population: 4168 CGM-glucometer matched data points analyzed, 67% of which were collected from the HG (ACCU-CHEK®). A total of 1375 matched data points were collected from the participants in the outpatient setting using the SIG (Contour®). There were 1435 matched pairs before radiation exposure and 2,733 matched data points after radiation exposure. Absolute blood glucose readings were plotted and analyzed using the Clarke Error Grid Analysis. Data points are matched blood glucose readings.
Measure: Count of Units; unit: Matched blood glucose readings
Units Other Than Participants: Matched blood glucose readings
Groups:
- CGM Uncovered -Pre Radiation Exposures: Uncovered CGM during radiologic procedures: Dexcom G6 CGM will not be covered during radiologic procedures, This data grouping provides baseline data.
- CGM Uncovered - Post Radiation Exposure: blood glucose readings after transmitter was exposed to scatter radiation.
- CGM Uncovered - Post Radiation Exposure >500 µGy: blood glucose readings after transmitter was exposed to scatter radiation greater than 500 µGy
- Handheld Clinical Glucometer: ACCU-CHEK handheld glucometer used in clinical setting
- Handheld Home Glucometer.: Contour glucometer used at home.
Arm/Group | CGM Uncovered -Pre Radiation Exposures | CGM Uncovered - Post Radiation Exposure | CGM Uncovered - Post Radiation Exposure >500 µGy | Handheld Clinical Glucometer | Handheld Home Glucometer.
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14
Number analyzed (Matched blood glucose readings) | 1435 | 1832 | 901 | 2793 | 1375
Matched blood glucose readings
  error grid section A | 806 | 1226 | 704 | 1715 | 1020
  error grid section B | 606 | 570 | 187 | 1033 | 329
  error grid section C | 6 | 7 | 5 | 56 | 69
  error grid section D | 17 | 31 | 5 | 47 | 15
Statistical Analysis 1: Comparison: CGM Uncovered -Pre Radiation Exposures vs CGM Uncovered - Post Radiation Exposure vs CGM Uncovered - Post Radiation Exposure >500 µGy vs Handheld Clinical Glucometer vs Handheld Home Glucometer; Test type: Other — Clarke error grid analyses (EGA) were performed to compare CGM values to glucometer glucose values blood glucose readings (mg/dL) were grouped based on radiation exposure (>0-500 µGy and >500 µGy). A p-value <0.05 was considered statistically significant; p < 0.05, Mixed Models Analysis; Generalized linear mixed models with random effects were used to assess absolute differences in BG mg/dL by cumulative scatter

2. Primary Outcome: Post Radiation Dexcom G6 Transmitter Functional Duration by Clark Error Analysis (Zone A and B %)
Description: Transmitter functional duration is determined by time from TPIAT procedure and CGM placement (baseline) to time for Transmitter changed (approximately 3 months), Functionality is determined by analysis of Blood Glucose (mg/dL) in month groupings (0-1month, 1-2months, 2+ months from baseline. Blood Glucose levels (mg/dL) obtained by the Dexcom G6 sensor and transmitter compared to blood glucose levels (mg/dL) obtained by a handheld glucometer until the transmitter is changed. The Clarke Error Grid Analysis method was used to compare absolute values. Accuracy reported as percentage of comparators in Zone A and B.
Time Frame: 3 months
Population: Data collected on functionality of transmitter over time (blood glucose (BG) mg/dL/months from TPIAT). Data points analyzed using the Clarke Error Grid analysis of matched blood glucose readings.
Measure: Count of Units; unit: Matched blood glucose readings
Units Other Than Participants: Matched blood glucose readings
Groups:
- Uncovered - 0-1 Month Post TPIAT: Transmitter matched data points (BG mg/dL) from 0-1 month post TPIAT
- Uncovered - 1-2 Months Post TPIAT: Transmitter matched data points (BG mg/dL) from 1-2months post TPIAT
- Uncovered - 2+ Months Post TPIAT: Transmitter matched data points (BG mg/dL) after 2 months post TPIAT
Arm/Group | Uncovered - 0-1 Month Post TPIAT | Uncovered - 1-2 Months Post TPIAT | Uncovered - 2+ Months Post TPIAT
Number analyzed (Participants) | 14 | 14 | 14
Number analyzed (Matched blood glucose readings) | 3294 | 586 | 288
Matched blood glucose readings
  error grid Zone A | 2065 | 446 | 226
  error grid Zone B | 1173 | 128 | 61
  error grid Zone C | 16 | 2 | 0
  error grid Zone D | 43 | 10 | 1
Statistical Analysis 1: Comparison: Uncovered - 0-1 Month Post TPIAT; Test type: Other — Clarke error grid analyses (EGA) were performed to compare CGM values to glucometer glucose values. A p-value <0.05 was considered statistically significant; p < 0.05, Mixed Models Analysis; Generalized linear mixed models with random effects over time were used to assess absolute differences in BG mg/dL by time

ADVERSE EVENTS:
Time Frame: Bassline to end of transmitter use (~3 months)
Description: Standard AE definitions were used in this study. There was no more than minimal risk for participants because they are using both the test device and the standard of care glucometer. Any elevated or low blood sugars levels would be caught by the monitoring system in place and would be acted on for clinical care.
Arm/Group | Uncovered
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05607576/Prot_SAP_000.pdf